CLINICAL TRIAL: NCT04903431
Title: Assessing the Effectiveness of Self- and Clinician-administered Crisis Response Planning for Suicide Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Lauren Khazem, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020B0414-B
Record Dates: First submitted 2021-05-18; First posted 2021-05-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician-administered Crisis Response Plan (Active Comparator): Clinicians will administer the Crisis Response Plan to 75 military veterans.
  Interventions: Behavioral: Crisis Response Planning for Suicide Risk
- Self-administered Crisis Response Plan (Experimental): Participants will complete a self-guided version of the Crisis Response plan online.
  Interventions: Behavioral: Crisis Response Planning for Suicide Risk

INTERVENTIONS:
Behavioral: Crisis Response Planning for Suicide Risk — Crisis Response Planning is focused on creating personalized set of steps for individuals to follow in case of a crisis and includes individuals' personal warning signs of distress, behavioral coping strategies, reasons for living, social supports to contact, and contact information for professional services, including emergency services. Personalization of the Crisis Response Plan is encouraged, and individuals are instructed to handwrite each step of the Crisis Response Plan on an index card to review.

SUMMARY:
The aim of the current project is to compare the use and preliminary effectiveness of a self-administered version of the Crisis Response Plan (CRP) in decreasing suicidal/death ideation and distress and increasing positive affect when compared to a clinician-administered version of the protocol in a sample of 150 military Veterans experiencing current death or suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* US military veteran
* death or suicidal ideation/suicide attempt within the past month

Exclusion Criteria:

* non-Veteran status
* acute intoxication or active psychosis precluding provision of informed consent
* inability to communicate and comprehend English
* residence outside the United States
* lack of past-month death/suicide ideation or attempt
* lack of device connected to webcam or internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Suicide Visual Analog Scale scores from the previous daily assessment | Administered daily for eight consecutive days
  The Suicide Visual Analog Scale The S-VAS assesses "urge to kill myself" using a horizontal line with anchors on the left reflecting "none" (score: 0) and on the right reflecting "extreme" (score: 100). The S-VAS is initially presented with the indicator on the "none" position, and non-movement of the indicator is followed by a prompt to remind the participant to move the indicator, if relevant, to ensure response accuracy. Higher scores are indicative of greater severity

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire - 2 scores from the previous daily assessment | Administered daily for eight consecutive days
  The PHQ-2 is a 2-item measure of depression symptom severity adapted from the 9-item version of the PHQ (Kroenke & Spitzer, 2002). Item responses are scores on a Likert scale ranging from 0 to 3. Total scores range from 0 to 6, with higher scores indicating greater symptom severity.
Change in Positive and Negative Affect Schedule - Short Form scores from the previous daily assessment | Administered daily for eight consecutive days
  The Positive and Negative Affect Schedule - Short Form a 20-item validated self-report measure of state positive and negative affect. The measure contains two, 10-item subscales measuring positive and negative affect, respectively. Possible total scores for each subscale range from 10 to 50, with higher scores indicating greater state affect.
Change in Crisis Response Plan Use from the previous daily assessment | Administered daily for eight consecutive days
  - In order to assess whether CRP use after completion impacts suicide urges and affect, participants will be instructed to "Please list all dates and times that you used part or all of the Crisis Response Plan that you completed since you last completed this survey. (or since you completed your Crisis Response Plan if this is the first survey you will complete)" You may provide us with your best estimates of dates and times."

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04903431/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT04903431/ICF_001.pdf